CLINICAL TRIAL: NCT01278433
Title: Large Scale Safety Study of IMOVAX Polio in Selected Cities in China, an Observational Post Marketing Study
Brief Title: A Safety Study of IMOVAX Polio Vaccine in Selected Cities in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IPV34; UTN: U1111 1115 6566 (Other: WHO)
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Polio; Poliomyelitis
Keywords: Polio; Poliovirus; IMOVAX Polio™
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental): Participants receiving their first dose of polio vaccine
  Interventions: Biological: IMOVAX Polio™: Inactivated Poliomyelitis Vaccine

INTERVENTIONS:
Biological: IMOVAX Polio™: Inactivated Poliomyelitis Vaccine — 0.5 mL, Intramuscular
  Other Names: IMOVAX Polio™

SUMMARY:
The aim of the study is to collect post marketing safety data on IMOVAX Polio vaccine in China.

Objective:

To describe serious adverse events 30 days after each dose of IMOVAX Polio™ administered at 2, 3, and 4 months of age among infants living in the study cities of China.

DETAILED DESCRIPTION:
Each study participant will receive an IMOVAX Polio™ injections at 2, 3 and 4 months of age (total of 3 doses) and will be followed up for 30 days after each vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 2 months of age or older (60-89days) when receiving the first dose of polio vaccine.
* Subject's parent /legal representative showed willingness to complete the 3 primary doses fully using IMOVAX Polio according to the schedule. one injection at 2, 3, 4 months old respectively;
* Informed consent form obtained by the subject's parent/legal representative.
* Subject plan to live in the selected study sites for at least three months after inclusion.

Exclusion Criteria:

* Subject with a history of serious illness (i.e., hypersensitivity, seizure, convulsion, encephalopathy diseases, etc.)
* Acute medical illness with or without fever within the last 72 hours.
* Vaccination planned in the 4 weeks following any trial vaccination (except Diphtheria, Tetanus, Pertussis (DTP), Hib vaccine or Pneumo vaccine)
* Participation in another clinical trial at the same time.
* Contraindications to vaccination according to IMOVAX Polio™ leaflet.
* Subject plan to leave the study sites for at least three months after inclusion.

Ages: 60 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5007 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting serious adverse events and relationship to Imovax Polio vaccination. | Up to 30 days after each vaccination
  A serious adverse event is defined as any untoward medical occurrence that at any dose (including overdose) results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect, or is an important medical event.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur China
Locations (15):
- China (15):
  - Beijing, Beijing Municipality
  - Changsha
  - Chengdu
  - Chongqing
  - Hangzhou
  - Jinan
  - Kunming
  - Nanjing
  - Qingdao
  - Shenyang
  - Shenzhen
  - Tianjin
  - Wuhan
  - Xi'an
  - Zheng Zho

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com